CLINICAL TRIAL: NCT06965803
Title: Continuous Glucose Monitor (CGM) Discharge Program
Brief Title: This Study is to Evaluate Whether Receiving Education and Glucose Monitoring With the CGM Device Will Improve Patient-reported Outcomes by Improving Patient's Satisfaction and Quality of Life (QOL) With Glucose Monitoring Device.
Acronym: CGM QOL
Status: Not yet recruiting | Type: Observational
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Matthew Monterola, Associate Director, Clinical Support Programs, Cedars-Sinai Medical Center
Other Study IDs: STUDY00003936
Record Dates: First submitted 2025-05-02; First posted 2025-05-11 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of the study is to improve patient-reported outcomes by improving patient's satisfaction and quality of life (QOL) with glucose monitoring device through pre and post satisfaction survey of patient with diabetes.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 or older
* diagnosed with Type 1 or Type 2 Diabetes who are on insulin
* able to speak and understand English language
* scheduled to receive a standard inpatient diabetes education consultation
* must not have used CGM in the six months prior to admission
* owns a smartphone
* demonstrates the ability to follow instructions and be capable of providing informed consent to participate in the program

Exclusion Criteria:

* those who are known to be pregnant. This is due to complexity of pregnancy-related changes in glucose metabolism and increased skin sensitivity, or changes in skin condition to adhesives and materials used in CGM devices.
* non-English speakers. As this is small study to evaluate which method is favorable using a survey only validated in English, enrolling non-English speakers would require additional resources/translations/personnel for evaluation and the education intervention that are not logistically possible right now.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: • Admitted patient with Type 1 or Type 2 diabetes.
Sampling Method: Non-Probability Sample
Enrollment: 37 (Estimated)
Dates: Start 2025-05-20 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Patient Satisfaction | 15 days
  Glucose Monitoring Satisfaction Survey

IPD SHARING:
Plan to Share IPD: No